CLINICAL TRIAL: NCT00168064
Title: A Phase II Pivotal Trial to Evaluate the Safety and Efficacy of Nitrogen Mustard (NM) 0.02% Ointment Formulations in Patients With Stage I or IIA Mycosis Fungoides (MF)
Brief Title: Safety and Efficacy of Nitrogen Mustard in Treatment of Mycosis Fungoides
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yaupon Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2005NMMF-201-US
Record Dates: First submitted 2005-09-07; First posted 2005-09-14 (Estimated); Results first posted 2012-10-31 (Estimated); Last update posted 2012-10-31 (Estimated); Status verified 2012-10

CONDITIONS: Mycosis Fungoides
Keywords: Mycosis Fungoides; Nitrogen Mustard; Cutaneous T-Cell Lymphoma; CTCL - Mycosis Fungoides
MeSH Terms: conditions — Mycosis Fungoides; Lymphoma, T-Cell, Cutaneous | interventions — Mechlorethamine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (PG - NM (MCH) 0.02%) (Active Comparator): PG - mechlorethamine-MCH (nitrogen mustard) 0.02% gel To evaluate the tolerability and safety of topical mechlorethamine-MCH (nitrogen mustard) 0.02% ointment formulations in patients with stage I or IIA MF
  Interventions: Drug: mechlorethamine-MCH (nitrogen mustard)
- 2 (AP - MCH(NM) 0.02%) (Active Comparator): AP - mechlorethamine-MCH (nitrogen mustard) 0.02% compounded in Aquaphor To evaluate the tolerability and safety of mechlorethamine-MCH (nitrogen mustard)0.02% ointment formulations in patients with stage I or IIA MF
  Interventions: Drug: mechlorethamine-MCH (nitrogen mustard)

INTERVENTIONS:
Drug: mechlorethamine-MCH (nitrogen mustard) — All affected areas (lesions) are to be treated once daily for twelve months with mechlorethamine-MCH (nitrogen mustard) 0.02% PG or NM 0.02% AP ointment
  Other Names: mechlorethamine; nitrogen mustard

SUMMARY:
This study will evaluate the efficacy, tolerability and safety of the topical application of mechlorethamine (MCH) formulations in patients with stage I or IIA mycosis fungoides (MF).

DETAILED DESCRIPTION:
The successful use of mechlorethamine (MCH) as a topical agent in the treatment of mycosis fungoides, a form of cutaneous T-cell lymphoma, was first reported in the late 1950s, and provided a rationale for skin-directed chemotherapy that minimized systemic toxicity. Since then, multiple investigators have demonstrated the safety and efficacy of topically applied MCH in the treatment of mycosis fungoides. This study will evaluate the efficacy (non-inferiority), tolerability and safety of topical application of MCH proprietary gel versus a compounded ointment formulation in Aquaphor in patients with stage I or IIA MF.

ELIGIBILITY:
Inclusion Criteria:

* Patients with mycosis fungoides confirmed by a skin biopsy
* Stage I or IIA patients must have been treated previously with prior topical therapies including PUVA, UVB, topical steroids, but not NM within the past 2 years, or topical carmustine (BCNU)
* Patients must be otherwise healthy with acceptable organ function.
* Prior to initiating study therapy, patients must not have had topical therapy within four weeks
* Lab values within normal range
* Willing/able to give consent
* Must use effective means of contraception if of childbearing potential

Exclusion Criteria:

* Newly diagnosed mycosis fungoides with no prior therapy
* A prior history of treatment with topical NM within the past 2 years or topical carmustine (BCNU)
* Use of topical or systemic therapies for MF within four (4) weeks of entry in the study
* Patients with a diagnosis of stage IIB-IV MF
* Serious known concurrent medical illness or infection, which could potentially present a safety risk and/or prevent compliance with the requirements of the treatment program
* Pregnant or nursing females, or males and females of childbearing potential, not using an effective means of contraception
* Patients who have had radiation therapy within one year of study start
* Patients who have a history of a higher T score than T2 or a higher N score than N1
* Patients who do not agree to do all labs at one site

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 260 (Actual)
Dates: Start 2006-05; Primary Completion 2010-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Lessin, M.D., Study Director — Fox Chase Cancer Center
Locations (12):
- United States (12):
  - Stanford University Medical Center, Stanford, California
  - Northwestern University - Dept. of Dermatology, Chicago, Illinois
  - NYU Medical Center Dept. of Dermatology, New York, New York
  - Columbia University, Dept. of Dermatology, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Oklahoma University, Tulsa, Oklahoma
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - University of Texas, Southwestern Medical Center, Dallas, Texas
  - The University of Texas, M.D. Anderson Cancer Center, Houston, Texas
  - Utah Clinical Trials, LLC, Salt Lake City, Utah
  - University of Wisconsin, Madison, Wisconsin

REFERENCES:
- [Background] Kim YH, Martinez G, Varghese A, Hoppe RT. Topical nitrogen mustard in the management of mycosis fungoides: update of the Stanford experience. Arch Dermatol. 2003 Feb;139(2):165-73. doi: 10.1001/archderm.139.2.165. PMID 12588222
- [Background] Kim YH. Management with topical nitrogen mustard in mycosis fungoides. Dermatol Ther. 2003;16(4):288-98. doi: 10.1111/j.1396-0296.2003.01640.x. PMID 14686971
- [Background] Kim YH, Jensen RA, Watanabe GL, Varghese A, Hoppe RT. Clinical stage IA (limited patch and plaque) mycosis fungoides. A long-term outcome analysis. Arch Dermatol. 1996 Nov;132(11):1309-13. PMID 8915308
- [Derived] Geskin LJ, Angello JT, Bagot M, Guenova E, Nikbakht N, Querfeld C, Scarisbrick JJ. Evaluating Response Trends of Chlormethine/Mechlorethamine Gel in Patients With Stage I-IIA Mycosis Fungoides: Analysis of Individual Patient Data From a Randomized Controlled Phase II Study to Facilitate Optimal Treatment Experiences. Clin Lymphoma Myeloma Leuk. 2024 Jan;24(1):40-47. doi: 10.1016/j.clml.2023.08.020. Epub 2023 Sep 7. PMID 37802679
- [Derived] Querfeld C, Scarisbrick JJ, Assaf C, Kim YH, Guitart J, Quaglino P, Hodak E. Chlormethine Gel Versus Chlormethine Ointment for Treatment of Patients with Mycosis Fungoides: A Post-Hoc Analysis of Clinical Trial Data. Am J Clin Dermatol. 2022 Jul;23(4):561-570. doi: 10.1007/s40257-022-00687-y. Epub 2022 May 10. PMID 35536441
- [Derived] Querfeld C, Scarisbrick JJ, Assaf C, Guenova E, Bagot M, Ortiz-Romero PL, Quaglino P, Bonizzoni E, Hodak E. Post hoc Analysis of a Randomized, Controlled, Phase 2 Study to Assess Response Rates with Chlormethine/Mechlorethamine Gel in Patients with Stage IA-IIA Mycosis Fungoides. Dermatology. 2022;238(2):347-357. doi: 10.1159/000516138. Epub 2021 Jun 4. PMID 34091453
- [Derived] Lessin SR, Duvic M, Guitart J, Pandya AG, Strober BE, Olsen EA, Hull CM, Knobler EH, Rook AH, Kim EJ, Naylor MF, Adelson DM, Kimball AB, Wood GS, Sundram U, Wu H, Kim YH. Topical chemotherapy in cutaneous T-cell lymphoma: positive results of a randomized, controlled, multicenter trial testing the efficacy and safety of a novel mechlorethamine, 0.02%, gel in mycosis fungoides. JAMA Dermatol. 2013 Jan;149(1):25-32. doi: 10.1001/2013.jamadermatol.541. PMID 23069814

RESULTS

PARTICIPANT FLOW:
Groups:
- PG -Mechlorethamine (Nitrogen Mustard) 0.02% PG Gel: Study formulation of Mechlorethamine-MCH (Nitrogen Mustard) 0.02% Gel
- AP- Mechlorethamine 0.02% Compounded in Aquaphor: Compounded Mechlorethamine-MCH (Nitrogen Mustard) in Aquaphor 0.02%
Period: Overall Study
Arm/Group | PG -Mechlorethamine (Nitrogen Mustard) 0.02% PG Gel | AP- Mechlorethamine 0.02% Compounded in Aquaphor
Started | 130 (128 participants received PG formulation) | 130 (127 participants received AP formulation)
Completed | 81 | 86
Not Completed | 49 | 44
Not completed — Adverse Event | 26 | 22
Not completed — Withdrawal by Subject | 3 | 4
Not completed — Lack of Efficacy | 4 | 4
Not completed — Lost to Follow-up | 4 | 3
Not completed — Non-compliance | 2 | 3
Not completed — Concurrent Illness | 4 | 3
Not completed — Subject's Best interest | 2 | 2
Not completed — Various | 4 | 3

BASELINE CHARACTERISTICS:
Groups:
- PG -Mechlorethamine-MCH (Nitrogen Mustard) 0.02% PG Gel: Study formulation of mechlorethamine-MCH (Nitrogen Mustard) 0.02% Gel
- AP- Mechlorethamine-MCH (NM) 0.02% Compounded in Aquaphor: Compounded mechlorethamine-MCH (Nitrogen Mustard)in Aquaphor 0.02%
- Total: Total of all reporting groups
Arm/Group | PG -Mechlorethamine-MCH (Nitrogen Mustard) 0.02% PG Gel | AP- Mechlorethamine-MCH (NM) 0.02% Compounded in Aquaphor | Total
Number analyzed (Participants) | 130 | 130 | 260
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 1 | 1
  Between 18 and 65 years | 93 | 86 | 179
  >=65 years | 37 | 43 | 80
Age Continuous [Mean (Standard Deviation); unit: years] | 54.7 (14.20) | 56.7 (14.34) | 55.7 (14.28)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53 | 53 | 106
  Male | 77 | 77 | 154
Region of Enrollment [Number; unit: participants]
  United States | 130 | 130 | 260

OUTCOME MEASURES:

1. Primary Outcome: Ratio of Response Rates Based on CAILS
Description: The ratio of the response rate of the patients treated with the PG formulation to the response rate of the patients treated with the AP formulation. Skin response determined by at least a 50% reduction from baseline in the Composite Assessment of Index Lesion Severity (CAILS) following up to 12 months of treatment
Time Frame: Assessment made at Day 1 and every subsequent visit during treatment
Population: ITT
Measure: Number; unit: percentage of participants
Groups:
- PG- Mechlorethamine-MCH (Nitrogen Mustard) 0.02% Gel: Study formulation of mechlorethamine-MCH (Nitrogen Mustard) 0.02% Gel
- AP- Aquaphor Formulation Mechlorethamine-MCH (NM) 0.02%: Mechlorethamine-MCH (Nitrogen Mustard) compounded in Aquaphor 0.02%
Arm/Group | PG- Mechlorethamine-MCH (Nitrogen Mustard) 0.02% Gel | AP- Aquaphor Formulation Mechlorethamine-MCH (NM) 0.02%
Number analyzed (Participants) | 130 | 130
percentage of participants | 76 | 62
Statistical Analysis 1: Comparison: PG- Mechlorethamine-MCH (Nitrogen Mustard) 0.02% Gel vs AP- Aquaphor Formulation Mechlorethamine-MCH (NM) 0.02%; Test type: Non-Inferiority or Equivalence — The PG formulation was determined to be non-inferior to the AP formulation if the lower limit of the 95% confidence interval around the ratio of the response rates (PG/AP) was > = 0.75; ANCOVA; ratio of proportions = 1.226, 95% CI 2-sided [0.974 to 1.552] — ratio is response rate of PG formulation divided by response rate of AP formulation

2. Secondary Outcome: Severity-weighted Assessment Tool (SWAT) Within up to 12 Months by 2 or More Consecutive Observations Over at Least 4 Weeks
Time Frame: Assessment made at Day 1 and every subsequent visit during treatment
Reporting Status: Not Posted

3. Secondary Outcome: Percent of Participants Achieving at Least 50% Improvement of Severity Weighted Assessment Tool (SWAT)
Description: Assessment of lesion distribution and severity. A responder analysis was performed on whether subject achieved at least 50% improvement on scale. This had to be confirmed on at least one visit at least 4 weeks apart.
Time Frame: Baseline to end of therapy
Measure: Number; unit: Percent of participants
Groups:
- AP- Mechlorethamine-MCH (NM) 0.02% Compounded in Aquaphor: Compounded mechlorethamine-MCH (Nitrogen Mustard) in Aquaphor 0.02%
Arm/Group | PG -Mechlorethamine-MCH (Nitrogen Mustard) 0.02% PG Gel | AP- Mechlorethamine-MCH (NM) 0.02% Compounded in Aquaphor
Number analyzed (Participants) | 130 | 130
Percent of participants | 61 | 60

ADVERSE EVENTS:
Time Frame: adverse event data were collected over 12 months of the patient's participation
Description: There were a total of 130 participants randomized to each treatment arm. However, 2 from the PG group and 3 from the AP group did not receive drug and are not included in the safety population.
Arm/Group | PG -Mechlorethamine-MCH (Nitrogen Mustard) 0.02% PG Gel | AP- Mechlorethamine-MCH (NM) 0.02% Compounded in Aquaphor
Serious Adverse Events (participants affected / at risk) | 0/128 | 0/127
Other Adverse Events (participants affected / at risk) | 108/128 | 99/127
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PG -Mechlorethamine-MCH (Nitrogen Mustard) 0.02% PG Gel (N=128) | AP- Mechlorethamine-MCH (NM) 0.02% Compounded in Aquaphor (N=127)
skin irritation (Skin and subcutaneous tissue disorders) | 32 (32) | 18 (18)
pruritus (Skin and subcutaneous tissue disorders) | 25 (25) | 20 (20)
erythema (Skin and subcutaneous tissue disorders) | 22 (22) | 18 (18)
dermatitis contact (Skin and subcutaneous tissue disorders) | 19 (19) | 19 (19)
skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 7 (7) | 9 (9)
upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 11 (11) | 10 (10)
folliculitis (Infections and infestations) | 7 (7) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No